CLINICAL TRIAL: NCT01497756
Title: Feasibility Trial of the Circumferential Abdominal Pelvic Pressure Device (CAPP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Mark Hauswald, Professor, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10-229
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Results first posted 2012-09-17 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CAPP application (Experimental): Patients in whom device is used
  Interventions: Device: CAPP use

INTERVENTIONS:
Device: CAPP use — Any abdominal pelvic pressure

SUMMARY:
A group of midwives and obstetric nurses have been trained to use circumferential abdominal pelvic pressure (CAPP) to treat postpartum hemorrhage. As part of the training follow up any use of a CAPP device will be monitored to identify complications.

DETAILED DESCRIPTION:
Providers will be surveyed twice at 4 and 8 months using open ended methods.

ELIGIBILITY:
Inclusion Criteria:

* Any patient receiving CAPP during study period.

Exclusion Criteria:

* None (CAPP is only clinically indicated for obstetric hemorrhage post delivery.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hauswald, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CAPP Application
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CAPP Application
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | NA — DOB was not solicited. All subjects were legal adults and in emergency situations.
  Between 18 and 65 years | NA — DOB was not solicited. All subjects were legal adults and in emergency situations.
  >=65 years | NA — No subjects were 65 or older since such patients are unable to become pregnant.
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — DOB was not solicited. All subjects were legal adults and in emergency situations.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Usage
Description: Number of patients on whom CAPP is used
Time Frame: Eight months
Population: Entire number of participants
Measure: Number; unit: participants
Arm/Group | CAPP Application
Number analyzed (Participants) | 10
participants | 10

2. Secondary Outcome: Side Effects
Description: Any recorded complications
Time Frame: Eight months
Population: All patients
Measure: Number; unit: participants
Arm/Group | CAPP Application
Number analyzed (Participants) | 10
participants | 0

ADVERSE EVENTS:
Arm/Group | CAPP Application
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes